CLINICAL TRIAL: NCT01992783
Title: The Effect of Resistant Starch Supplementation on Antioxidant Status and Insulin Resistance in Overweight and Obese Adults
Brief Title: Resistant Starch, Antioxidant Status and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: umsu.rec.1392.75
Record Dates: First submitted 2013-11-05; First posted 2013-11-25 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Overweight; Obesity
Keywords: Resistant Starch; Antioxidant Status; Insulin Resistance; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — high-amylose maize type 2 resistant starch, maize; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hi-maize resistant starch (Experimental): 13.5 g/day
  Interventions: Dietary Supplement: Hi-maize resistant starch
- Maltodextrin (Placebo Comparator): 13.5 g/day
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Hi-maize resistant starch — 13.5 g/day
  Arms: Hi-maize resistant starch
Dietary Supplement: Maltodextrin — 13.5 g/day
  Arms: Maltodextrin

SUMMARY:
The aim of this study is to evaluate whether supplementation with resistant starch improves biomarkers associated with antioxidant status and insulin resistance in subjects with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adults
* Age: 20-50 years

Exclusion Criteria:

* weight loss or gain (more than10%) over the past 6 months, or weight loss (more than 5%) over the past 1 month
* pregnancy, lactation or menopause
* History of acute disease or clinical evidence of cancer, acute or chronic inflammatory diseases, cardiovascular disease, renal disease, liver disease, thyroid or endocrine disease
* Gastrointestinal disease of which ingredients found in the study products have adverse effects on that
* Use of antihypertensive, lipid lowering or glucose lowering medications
* Taking antioxidant, vitamin, and/or mineral supplements
* smoking

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Antioxidant status | 4 weeks
  Superoxide dismutase (SOD), Plasma malondialdehyde (MDA), Total antioxidant capacity (TAC)

SECONDARY OUTCOMES:
Insulin resistance | 4 weeks
  Fasting glucose, Fasting insulin, Insulin resistant (HOMA-IR)
Lipid profile | 4 weeks
  Triglyceride, Total cholesterol, HDL-cholesterol, LDL-cholesterol, Total cholesterol/HDL-cholesterol
Blood pressure | 4 weeks
Anthropometric parameters | 4 weeks
  Height, Weight, Body Mass Index (BMI), Waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alizadeh, PhD, Principal Investigator — Assistant Professor in Nutrition
Locations (1):
- Urmia, Azerbaijan-gharbi, Iran

REFERENCES:
- [Derived] Eshghi F, Bakhshimoghaddam F, Rasmi Y, Alizadeh M. Effects of Resistant Starch Supplementation on Glucose Metabolism, Lipid Profile, Lipid Peroxidation Marker, and Oxidative Stress in Overweight and Obese Adults: Randomized, Double-Blind, Crossover Trial. Clin Nutr Res. 2019 Oct 28;8(4):318-328. doi: 10.7762/cnr.2019.8.4.318. eCollection 2019 Oct. PMID 31720257